CLINICAL TRIAL: NCT02074020
Title: A Randomized, Double-Blind, Placebo-Controlled Phase 3 Study to Evaluate the Efficacy and Safety of Blisibimod Administration in Subjects With Systemic Lupus Erythematosus With or Without Nephritis
Brief Title: CHABLIS-SC2: A Study of the Efficacy and Safety of Subcutaneous Blisibimod in Subjects With Systemic Lupus Erythematosus With or Without Nephritis
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Anthera Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AN-SLE3332
Record Dates: First submitted 2014-02-26; First posted 2014-02-28 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2015-08

CONDITIONS: Systemic Lupus Erythematosus
Keywords: SLE; Lupus; Lupus Erythematosus, Systemic; Autoimmune Diseases; A-623; Blisibimod; Nephritis
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Autoimmune Diseases; Nephritis | interventions — AMG623 peptibody

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Blisibimod (Experimental)
  Interventions: Drug: Blisibimod
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Blisibimod — Administered via subcutaneous injection once per week
  Arms: Blisibimod
Drug: Placebo — Administered via subcutaneous injection once per week
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the clinical efficacy of blisibimod as measured by a composite responder index in subjects who, despite corticosteroid use, continue to have autoantibody positive, clinically-active Systemic Lupus Erythematosus (SLE) as defined by SELENA SLEDAI score ≥10.

ELIGIBILITY:
Inclusion Criteria:

* Fulfill at least 4 diagnostic criteria for SLE defined by American College of Rheumatology
* Positive antinuclear antibodies (ANA) and/or anti-double stranded DNA (anti-dsDNA)
* Active SLE disease as defined by SELENA-SLEDAI score ≥10 despite on-going stable corticosteroid therapy
* Subjects with stable nephritis may be enrolled
* 18 years of age or older

Exclusion Criteria:

* Severe active vasculitis, active central nervous system lupus, uncontrolled hypertension or poorly controlled diabetes
* Malignancy within past 5 years
* Known to be positive for HIV and/or positive at the screening visit for hepatitis B, or hepatitis C
* Liver disease
* Anemia, neutropenia, or thrombocytopenia
* Active infection requiring hospitalization or treatment with parenteral antibiotics within the past 60 days or history of repeated herpetic viral infections
* History of active tuberculosis or a history of tuberculosis infection
* Pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-12; Primary Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Proportion of responders to the SRI-8 composite responder index | 52 Weeks

SECONDARY OUTCOMES:
Time to first severe SLE flare | Baseline through 52 weeks
Change in the number of actively tender or swollen joints and in mucocutaneous disease activity | 52 Weeks
Change in proteinuria from baseline | Week 52
Proportion of subjects able to reduce oral steroid dose | Baseline through 52 weeks
Proportion of subjects with improved patient-reported outcomes | Week 52
Time to treatment failure | Through week 52
Change from baseline in B cell subsets, anti-dsDNA, C3, C4 | Through week 52
Safety profile (AEs, vital signs, labs, physical exams) | Through week 52

OTHER OUTCOMES:
Subgroup analyses of blisibimod effect in subjects with renal manifestations at baseline | 52 Weeks

REFERENCES:
- [Derived] Hannon CW, McCourt C, Lima HC, Chen S, Bennett C. Interventions for cutaneous disease in systemic lupus erythematosus. Cochrane Database Syst Rev. 2021 Mar 9;3(3):CD007478. doi: 10.1002/14651858.CD007478.pub2. PMID 33687069